CLINICAL TRIAL: NCT01981720
Title: A Multi Center Extension Study of PRX-102 Administered by Intravenous Infusions Every 2 Weeks for up to 60 Months to Adult Fabry Patients
Brief Title: Extension Study of PRX-102 for up to 60 Months
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Protalix (Industry)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-102-F03
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Results first posted 2023-02-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Fabry Disease
Keywords: PRX-102; pegunigalsidase alfa; Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- PRX-102 (pegunigalsidase alfa) (Experimental): PRX-102 (pegunigalsidase alfa) 1.0 mg/kg IV every 2 weeks (+/- 3 days)
  Interventions: Biological: PRX-102 (pegunigalsidase alfa)

INTERVENTIONS:
Biological: PRX-102 (pegunigalsidase alfa) — PRX-102 1 mg/kg every 2 weeks
  Other Names: pegunigalsidase alfa; Recombinant human alpha galactosidase-A

SUMMARY:
To evaluate the ongoing safety, tolerability, and efficacy parameters of PRX-102 in adult Fabry patients who have successfully completed treatment with PRX-102 in studies PB-102-F01 and PB-102-F02.

DETAILED DESCRIPTION:
An open-label study to evaluate the ongoing safety, tolerability and efficacy parameters of PRX-102 in adult Fabry patients (≥18 years of age). Patients enrolled received 1.0 mg/kg of PRX-102 as an intravenous infusion every 2 weeks (+/- 3 days) for up to 60 months and no less than 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Completion of study PB-102-F02
* The patient signs informed consent
* Female patients and male patients whose co-partners were of child-bearing potential agree to use a medically acceptable method of contraception, not including the rhythm method. Acceptable methods of contraception include hormonal products, intrauterine device, or male or female condoms. Contraception should be used throughout the duration of the study and for 3 months after termination of treatment.

Exclusion Criteria:

* Presence of any medical, emotional, behavioral or psychological condition that, in the judgment of the Investigator and/or Medical Director, would interfere with the patient's compliance with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01-16 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2021-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - University of Florida, Gainesville, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Institute of Metabolic Disease, Dallas, Texas
  - O & O Alpan, Fairfax, Virginia
- Instituto Privado de Hematologia E Investigacion Clinica (I.P.H.I.C), Asunción, Paraguay
- Hospital de Dia Quiron Zaragoza, Zaragoza, Spain
- The Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult Fabry disease patients who have successfully completed treatment with PRX-102 in previous studies PB-102-F01 and PB-102-F02
Pre-assignment Details: A total of 15 adult patients (8 male and 7 female) who completed study PB-102-F02 were enrolled in this study and included in both the Safety and Efficacy populations.
Period: Overall Study
Arm/Group | PRX-102 (Pegunigalsidase Alfa)
Started | 15
Completed | 10
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | PRX-102 (Pegunigalsidase Alfa)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11
  United Kingdom | 1
  Paraguay | 1
  Spain | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.03
Description: Results represent the number of treatment-emergent adverse events (TEAE) that were considered definitely, probably or possibly related to study treatment.
Time Frame: Every two weeks up to 60 months
Population: Safety population is defined as all patients who received any dose (partial or complete) of study treatment as part of study PB-102-F03. Efficacy population is defined as all patients who received at least one complete dose of the study treatment as part of study PB-102-F03
Measure: Number; unit: participants
Arm/Group | PRX-102 (Pegunigalsidase Alfa)
Number analyzed (Participants) | 15
participants
  Safety Analysis Set : At lease 1 TEAE | 13
  Safety Analysis Set : At least 1 mild or moderate TEAE | 13
  Safety Analysis Set : At least 1 severe TEAE | 5
  Safety Analysis Set : At least 1 SAE | 2
  Safety Analysis Set : At least 1 definitely, probably or possibly related | 4
  Safety Analysis Set : At least 1 TEAE leading to discontinuation | 1
  Safety Analysis Set : At least 1 TEAE leading to death | 1

2. Other Pre Specified Outcome: Plasma Lyso-Gb3 Concentration
Description: Globotriaosylsphingosine (Lyso-Gb3) is Fabry disease specific biomarker, which was measured at Baseline, every 3 months up to 24 months and then every 6 months up to the end of the study. Baseline and Month 60 and change from Baseline reported.
Time Frame: Baseline and month 60
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Efficacy Population: All patients who received at least one complete dose of the study treatment as part of study PB-102-F03
- Male; Female: Subject analysis set
Arm/Group | Efficacy Population | Male | Female
Number analyzed (Participants) | 15 | 8 | 7
ng/mL
  Baseline | 70.8 (20.4) | 124.4 (25.9) | 9.6 (2.1)
  Month 60 | 6.4 (1.5) | 9.2 (1.6) | 2.1 (0.9)
  Change from Baseline to Month 60 | -68.4 (25) | -111.0 (31) | -4.6 (0.9)

3. Other Pre Specified Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR was calculated based on the serum creatinine values according to the CKD-EPI equation. The absolute change in eGFR from baseline measurement at visit 1 to Month 60 was summarized using descriptive statistics. Baseline and month 60 reported.
Time Frame: Baseline and Month 60
Measure: Mean (Standard Error); unit: ml/min/1.73 m^2
Groups:
- Efficacy Population; Male; Female: Subject analysis set
Arm/Group | Efficacy Population | Male | Female
Number analyzed (Participants) | 15 | 8 | 7
ml/min/1.73 m^2
  Baseline | 111.7 (5.5) | 118.1 (7.7) | 104.45 (7.5)
  Month 60 | 97.0 (6.4) | 100.0 (8.3) | 92.4 (11.4)
  Change from Baseline to Month 60 | -10.9 (2.0) | -14.5 (1.7) | -5.6 (2.6)

ADVERSE EVENTS:
Time Frame: The adverse events were collected during the period from PB-102-F03 baseline up to the end of study PB-102-F03 (up to 60 months).
Arm/Group | PRX-102 (Pegunigalsidase Alfa)
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRX-102 (Pegunigalsidase Alfa) (N=15)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRX-102 (Pegunigalsidase Alfa) (N=15)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Chest pain (General disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (2)
Feeling hot (General disorders) | 1 (1)
Infusion site bruising (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 1 (1)
Pruritis genital (Reproductive system and breast disorders) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (3)
Cardiac murmur (Investigations) | 1 (1)
Abnormal chest x-ray (Investigations) | 1 (1)
Electrocardiogram ST segment abnormal (Investigations) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 1 (1)
Nuclear magnetic resonance imaging abnormal (Investigations) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus arrythmia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (3)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Ventricular hypertrophy (Cardiac disorders) | 1 (1)
Fabry's disease (Congenital, familial and genetic disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (12)
Paraesthesia (Nervous system disorders) | 4 (6)
Dizziness (Nervous system disorders) | 2 (3)
Balance disorder (Nervous system disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Visual field defect (Nervous system disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (3)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Deafness bilateral (Ear and labyrinth disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 4 (9)
Abdominal pain (Gastrointestinal disorders) | 4 (9)
Diarrhoea (Gastrointestinal disorders) | 4 (9)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Clubbing (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (8)
Upper respiratory tract infections (Infections and infestations) | 5 (8)
Influenza (Infections and infestations) | 3 (4)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (3)
Herpes virus infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (3)
Onychomycosis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (3)
Sinusitis (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (5)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial agreement provided to the sites and Investigators contains a Publication paragraph that indicates the following: shall not, without the Sponsor's prior written consent, independently publish, present or otherwise disclose any results of or information pertaining to the trial until a multicenter publication is published, subject to certain limitations regarding timing and the confidentiality of unpublished data.

DOCUMENTS (2):
  • Study Protocol (2016-01-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT01981720/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT01981720/SAP_001.pdf